CLINICAL TRIAL: NCT03218761
Title: Validation of Norepinephrine Transporter (NET) mRNA as a Measure of Functional NET Expression in Postural Tachycardia Syndrome (POTS)
Brief Title: POTS NET mRNA Functional Correlation With NET Activity
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Calgary (Other); Dysautonomia International (Other)
Responsible Party: Principal Investigator, Satish R. Raj, Adjunct Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: IRB#170714
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Postural Tachycardia Syndrome
Keywords: norepinephrine; norepinephrine transporter
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Plasma samples supine and upright catechol levels Urine for catechol levels PAXgene tubes for RNA assessment plasma/serum aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POTS Patients: Patients who self-identify as having Postural Tachycardia Syndrome.
  They will have assessment of NET mRNA levels, supine plasma catechols, standing plasma catechols, and urine catechols.
  Interventions: Diagnostic Test: NET mRNA level; Diagnostic Test: Plasma catechols; Diagnostic Test: Urine Catechols
- Control Subjects: Subjects who do not have Postural Tachycardia Syndrome.
  They will have assessment of NET mRNA levels, supine plasma catechols, standing plasma catechols, and urine catechols.
  Interventions: Diagnostic Test: NET mRNA level; Diagnostic Test: Plasma catechols; Diagnostic Test: Urine Catechols

INTERVENTIONS:
Diagnostic Test: NET mRNA level — quantification of mRNA to the Norepinephrine Transporter (NET)
Diagnostic Test: Plasma catechols — plasma for assay of norepinephrine (NE), DHPG (intraneuronal metabolite of NE), and other catechols
Diagnostic Test: Urine Catechols — urine for assay of norepinephrine (NE), DHPG (intraneuronal metabolite of NE), and other catechols

SUMMARY:
DNA Acetylation can be responsible for significant down-regulation of transcription of the Norepinephrine Transporter (NET). NET is an important clearance transporter that removes norepinephrine (NE) from sympathetic neuronal synapses. Very low levels of NET can "cause" Postural Tachycardia Syndrome (POTS) or make these patients more susceptible to certain medications. Quantified NET messenger RNA (mRNA) levels from a peripheral blood sample may be able to assess NET availability, which is simpler than older methods. This has not been validated against NET function. In this protocol, the investigators seek to assess whether these NET mRNA levels correlate with NET function. The investigators will assess the DHPG (NET dependent NE metabolite):NE ratio in POTS patients and control subjects from both plasma and urine samples.

DETAILED DESCRIPTION:
Work from The Baker Institute in Melbourne, Australia has shown that there can be significant epigenetic modification of the Norepinephrine Transporter (NET). DNA Acetylation can be responsible for significant down-regulation of transcription. NET is an important clearance transporter that removes norepinephrine (NE) from sympathetic neuronal synapses.Very low levels of NET can produce a hyperadrenergic phenotype and can "cause" Postural Tachycardia Syndrome (POTS). The Baker Institute researchers have started using quantified NET mRNA levels from a peripheral blood sample to assess NET availability. This is a huge advance due to its simplicity, in contrast to a prior method which involved a vein biopsy to look at the level of protein expression.

In this protocol, the investigators seek to assess whether these NET messenger RNA (mRNA) levels correlate with NET function. When NET transports NE back into presynaptic neurons, a high percentage gets converted to a metabolite (DHPG) and then released into the blood stream. Therefore, the ratio of DHPG:NE ratio is decreased with reduced NET activity. The investigators will assess this DHPG:NE ratio in POTS patients and control subjects from both plasma and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* • Postural Tachycardia Syndrome

  * Previously diagnosed with POTS

    • Control Subjects
  * Not diagnosed with POTS

    * Age between 13-80 years
    * Male and female subjects are eligible.
    * Able and willing to provide informed consent (if ≥18 years) or assent with parental consent (if age 13-17 years)

Exclusion Criteria:

* • Inability to give, or withdrawal of, informed consent

  * Use of serotonin-norepinephrine reuptake inhibitors (SNRI) or NET inhibitors within 1 month

    o These drugs pharmacologically block NET activity
  * Use of Tricyclic antidepressants within 1 week

    o Many tricyclic antidepressants pharmacologically block NET activity
  * Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with POTS and Subjects without POTS who are not on drugs that inhibit the norepinephrine transporter and are willing to give their informed consent (or assent and parental consent) to participate in the project.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-14 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Supine Plasma DHPG:NE correlation | 1 day
  NET mRNA above and below median supine plasma DHPG:NE

SECONDARY OUTCOMES:
Standing Plasma DHPG:NE correlation | 1 day
  NET mRNA above and below median standing plasma DHPG:NE
Urine DHPG:NE correlation | 1 day
  NET mRNA above and below median urine DHPG:NE

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No